CLINICAL TRIAL: NCT05540093
Title: Influence of Adding High Power Pain Threshold Ultrasound to Traditional Therapy on Axioappendicular Muscles Amplitude and Fatigue in Mechanical Neck Pain Randomized Clinical Trials
Acronym: MNP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: p.t.REC/012/003619
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Neck Pain
Keywords: high power pain threshold ultrasound; mechanical neck pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: high power pain threshold ultrasound and traditional therapy
Who Masked: Outcomes Assessor
Masking Description: permuted block randomization
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high power pain threshold ultrasound (Experimental): the patients will receive high power pain threshold ultrasound and traditional therapy twice a week for four weeks
  Interventions: Other: high power pain threshold ultrasound; Other: traditional therapy
- traditional therapy (Active Comparator): the patients will receive traditional therapy twice a week for four weeks
  Interventions: Other: traditional therapy

INTERVENTIONS:
Other: high power pain threshold ultrasound — After explaining the procedure, and the trigger points will be marked by a physical therapist that . Then, the hand placed next to the prone position with the head in the neutral position, and the hands placed next to the body. The frequency was set to 1 MHz, and the intensity increased from 0.5 to 2 until the patient reported an unpleasant sensation. The probe will be held there for 4 s; then, the intensity was reduced by 50%, and the probe was moved over and around the trigger point. This process is done several times for three minutes.
  Arms: high power pain threshold ultrasound
Other: traditional therapy — the patients will receive traditional therapy in the form of postural correction exercise, active range of motion and stretching exercise for cervical muscles

SUMMARY:
The purpose of this study will investigate the effect of adding high power pain threshold ultrasound to traditional therapy on axioappendicular muscles amplitude and fatigue in neck pain

DETAILED DESCRIPTION:
Myofascial pain syndrome is a common musculoskeletal pain disorder affecting almost 95% of people with chronic pain disorders and is a common finding in especially pain management centres.It is characterized by trigger points, defined as hyperirritable spots within taut bands of skeletal muscle fibers. The syndrome is associated with tenderness in the muscle, referred pain, spasm and restriction of motion. Patients with MPS begin with one active MTrP (called the primary MTrP) in the affected muscles due to chronic repetitive minor muscle strain, poor posture, systemic diseases, or neuro-musculoskeletal lesions. When not treated correctly, expansion of the pain region and additional active MTrPs (called secondary or satellite MTrPs) will develop one of the most appropriate treatments for trigger points ultrasound therapy. The high-power pain threshold ultrasound (HPPTUS) technique is one of the ultrasound modifications used to treat trigger points In 2004, Majlesi et al. performed the first clinical study to compare this technique with the traditional ultrasound technique in patients with myofascial trigger points. The results showed that HPPTUS was much more effective than the traditional technique, and pain reduction and improved range of motion (ROM) were significant in a smaller number of sessions.sixty patients with mechanical neck pain will be assigned randomly to two equal group. one group will receive high power pain threshold ultrasound and traditional therapy and the other receive traditional therapy alone for four weeks.

.

ELIGIBILITY:
Inclusion Criteria:

* patients with mechanical neck pain from both genders.
* age between 19 and 38 years
* patients will be required to have active TrPs in the upper trapezius and levator muscle and neck pain

Exclusion Criteria:

* Patients will be excluded if they have History of whiplash injury,
* History of cervical spine surgery,
* Cervical radiculopathy or myelopathy,
* Having undergone physical therapy within the past 3 months before the study
* Non- rheumatologic diseases as multiple sclerosis,
* thyroid dysfunction and chronic infection and Rheumatologic condition as mild systemic lupus erythematosus, poly-articular osteoarthritis, rheumatoid arthritis and advanced cervical spine degenerative diseases.

Ages: 19 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
pain intensity | up to four weeks
  pain will be measured by visual analogue scale
pressure pain threshold | up to four weeks
  commander algometer device will be used to measure pressure pain threshold

SECONDARY OUTCOMES:
neck disability | up to four weeks
  neck disability index will be used to measure neck disability.
muscle amplitude and fatigue | up to four weeks
  electromyography will be used to measure muscle amplitude and fatigue

CONTACTS AND LOCATIONS:
Locations (1):
- Al Shaymaa Shaaban Abd El Azeim, Giza, Egypt